CLINICAL TRIAL: NCT06531161
Title: Safety and Efficacy of Suxiao Jiuxin Pill for Prevention of Acute Mountain Sickness: a Randomized Controlled Trial
Brief Title: EleVation carE: a Randomized Controlled Trial on the Prevention of Acute Mountain Sickness With Suxiao Jiuxin Pill
Acronym: EVEREST
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Tibet Autonomous Region Hospital of Traditional Tibetan Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SXJX-AMS-02
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Acute Mountain Sickness
Keywords: Acute Mountain Sickness; Suxiao Jiuxin Pill; Traditional Chinese Medicine
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, care providers, investigators, and outcome assessors will be blinded throughout the clinical trial. To ensure blindness, the experimental drug and placebo will be similar in dosage, odor, and taste. Suxiao Jiuxin Pill and placebo will be repackaged and distributed according to standardized procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Suxiao Jiuxin Pill group (Experimental): Participants who are randomly assigned to Suxiao Jiuxin Pill group will receive Suxiao Jiuxin Pills (6 pills per time, 3 times a day, taken sublingually) for 4 days at sea level and another 3 days at high altitude.
  Interventions: Drug: Suxiao Jiuxin Pill
- Placebo: Placebo group (Placebo Comparator): Participants who are randomly assigned to Placebo group will receive placebo (6 pills per time, 3 times a day, taken sublingually) for 4 days at sea level and another 3 days at high altitude.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suxiao Jiuxin Pill — Suxiao Jiuxin Pill is a traditional Chinese medicine compound composed of Ligusticum Wallichii and Borneo Camphorwood, and its clinical safety has been confirmed. Traditional Chinese medicine theory believes that Suxiao Jiuxin Pill has the effects of promoting qi and blood circulation, removing blood stasis and relieving pain, which may help alleviate symptoms of AMS.
  Arms: Experimental: Suxiao Jiuxin Pill group
Drug: Placebo — Placebo is made of less than 10% of the amount of Suxiao Jiuxin Pill, with similar dosage, odor, and taste.
  Arms: Placebo: Placebo group

SUMMARY:
The aim of this randomized, controlled trial is to evaluate the safety and efficacy of Suxiao Jiuxin Pills for prevention of acute mountain sickness (AMS) after high altitude exposure in healthy volunteers, and its influences on physiological indicators before and after high altitude exposure.

DETAILED DESCRIPTION:
Acute altitude illness refers to a group of clinical symptoms that occur when travelers are exposed to high altitude in a short period of time, due to the body's incomplete or dysregulated adaptation to hypoxic environment, which may occur at anytime from a few hours to 5 days after ascending, with severity ranging from mild discomfort to life-threatening conditions such as cerebral and pulmonary edema. AMS is the most common manifestation, characterized by headache, gastrointestinal symptoms, fatigue, weakness, dizziness, light-headedness, etc. Lake Louise Score (LLS) system has been widely used to evaluate AMS, and the version updated in 2018 kept nausea/vomiting, fatigue, lassitude and dizziness as the assessment symptom for AMS, and each symptom can be scored as 0-3 according to severity. AMS can be diagnosed when headache exist and total LLS is ≥ 3 points. Based on total scores, AMS can be defined as mild (3-5), moderate (6-9) and severe (10-12).

Suxiao Jiuxin Pill is a traditional Chinese medicine compound composed of Ligusticum Wallichii and Borneo Camphorwood, and its clinical safety has been confirmed. A total of 168 subjects will be enrolled in this randomized, controlled trial, and eligible subjects will be randomized into Suxiao Jiuxin Pill intervention group or Placebo group after informed consent is obtained. The study drug or placebo will be given orally for 4 days at sea level, arrival day and another 2 days at high altitude. The clinical assessments, including LLS system, sleep questionnaire scores, vital signs, blood oxygen saturation, blood routine test, blood biochemistry test, echocardiogram, Holter, ambulatory blood pressure monitoring, pulse wave velocity, and transcranial Doppler ultrasound parameters will be repeatedly performed at sea level and high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged 18-55 years old (including boundary values);
* Female volunteers weighing ≥45.0 kg and male volunteers weighing ≥50.0 kg, with a body mass index (BMI) between 19.0 and 28.0 kg/m2 (including boundary values) (BMI=weight kg/height m2);
* Primary residence at an altitude of <500 meters above sea level;
* Not ascending to an altitude >2500 meters in the 6 months prior to the screening period;
* Voluntary participation with written informed consent.

Exclusion Criteria:

* Subjects with previous severe high altitude sickness such as high altitude heart disease, high altitude pulmonary edema, high altitude cerebral edema, and high altitude erythrocytosis;
* Subjects with established cardiovascular or cerebrovascular disease or uncontrolled hypertension (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg at screening);
* Subjects with clinically significant respiratory disease, digestive disease, liver disease, central nervous system disease, psychiatric disease, metabolic disease, renal disease, anemia, or acute infection;
* Subjects with primary headache (migraine, tension headache, cluster headache, etc.) or secondary headache (headache associated with infection, cerebrovascular, etc.) within 1 month prior to screening;
* Subjects with insomnia, anxiety, depression or a history of motion sickness or airplane sickness;
* Subjects with Lake Louise Score ≥ 2 at screening;
* Subjects with left index finger oxygen saturation <95% at screening;
* Subjects with alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of the normal range, or creatinine > upper limit of the normal range at screening;
* Subjects with hypersensitive C-reactive protein > upper limit of normal range at screening;
* Subjects with history of surgery or blood donation within 3 months prior to screening;
* Subjects with any medication or non-pharmacological intervention (including dietary supplements) to prevent or treat acute mountain sickness within 14 days prior to screening;
* Smoking ≥20 cigarettes per day within 3 months prior to screening;
* Contraindications to the use of Suxiao Jiuxin Pill, such as allergies;
* Women who are pregnant, breastfeeding, or have a positive pregnancy test (human chorionic gonadotropin test);
* Alcohol abuse [more than 28 standard units of alcohol per week (1 standard unit contains 14 g of alcohol, e.g., 360 mL of beer, 45 mL spirit with 40% alcohol by volume, or 150 mL of wine)] or substance abuse within 6 months prior to screening;
* Participation in another interventional clinical study within 3 months prior to screening;
* Other conditions, in the opinion of the investigators, make participation in this study inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of AMS assessed by LLS system on the next morning of arrival day at high altitude between Suxiao Jiuxin Pill and Placebo groups. | The next morning of arrival day at high altitude
  AMS was defined as LLS score ≥ 3 with headache and at least one of the symptoms of nausea or vomiting, fatigue, dizziness. The difference in incidence rate of AMS on the next morning of arrival day at high altitude is pre-specified as primary efficacy endpoint between Suxiao Jiuxin Pill and Placebo groups.

SECONDARY OUTCOMES:
Incidence rate of AMS assessed by LLS system after arrival at high altitude between Suxiao Jiuxin Pill and Placebo groups. | Arrival day to Day 3 after high altitude exposure
  LLS assessments will be conducted before breakfast and before sleep after arrival at high altitude. The difference will be compared in the total incidence rates of AMS assessed by LLS after arrival between Suxiao Jiuxin Pill and Placebo groups.
Baseline-corrected LLS after high altitude exposure between Suxiao Jiuxin Pill and Placebo groups. | Day 4 at sea level to Day 3 after high altitude exposure
  LLS assessments will be conducted before breakfast and before sleep on Day 4 (at sea level) and the days after high altitude exposure. LLS on Day 4 will be used as baseline scores. The difference will be compared in the mean baseline-corrected LLS between Suxiao Jiuxin Pill and Placebo groups.
Area under the curve (AUC) of LLS in the mean LLS score-time profile after arrival between Suxiao Jiuxin Pill and Placebo groups. | Arrival day to Day 3 after high altitude exposure
  LLS assessments will be conducted before breakfast and before sleep on days after arrival. The AUC of LLS in the mean LLS score-time profile after arrival will be compared between Suxiao Jiuxin Pill and Placebo groups.
Incidence rate of moderate and above AMS on the next morning of arrival at high altitude between Suxiao Jiuxin Pill and Placebo groups. | The next morning of arrival day at high altitude
  Moderate and above AMS is defined as LLS score ≥ 6. The difference will be compared in the incidence rates of moderate and above AMS on the next morning of arrival between Suxiao Jiuxin Pill and Placebo groups.
Mean AMS Clinical Functional Score after arrival between Suxiao Jiuxin Pill and Placebo groups. | Arrival day to Day 3 after high altitude exposure
  Self-reported AMS Clinical Functional Score is used to evaluate the impact of AMS symptoms on overall function at high altitude. The difference will be compared in the AMS Clinical Functional Scores after arrival between Suxiao Jiuxin Pill and Placebo groups.
Blood oxygen saturation (SpO2) from sea level to high altitude between Suxiao Jiuxin Pill and Placebo groups. | Day 4 at sea level to Day 3 after high altitude exposure
  Blood oxygen saturation (SpO2) will be tested using a pulse oximetry and measured from the left index finger. SpO2 will be tested for 3 times daily by staff before breakfast, before lunch, and before sleep from Day 4 at sea level to Day 3 after high altitude exposure. The difference will be compared in SpO2 from sea level to high altitude between Suxiao Jiuxin Pill and Placebo groups.
Incidence rate of AMS symptoms requiring additional treatment during and after high altitude exposure between Suxiao Jiuxin Pill and Placebo groups. | Arrival day to Day 3 after high altitude exposure
  AMS symptoms requiring additional treatment is defined as high-altitude cerebral edema, high-altitude pulmonary edema, and severe AMS symptoms (nausea, vomiting, fatigue, dizziness, etc.). The difference will be compared in the incidence rates of AMS symptoms requiring additional treatment during and after high altitude exposure between Suxiao Jiuxin Pill and Placebo groups.
Acute Mountain Sickness Symptom Scale and Score after arrival between Suxiao Jiuxin Pill and Placebo groups. | Arrival day to Day 3 after high altitude exposure
  Acute Mountain Sickness Symptom Scale and Score is a scoring system which evaluates symptoms of headache, vomiting, dizziness, nausea, palpitation, shortness of breath, chest tightness, dizziness, insomnia, drowsiness, loss of appetite, abdominal distention, diarrhea, constipation, cyanosis of the lips, numbness of the hands and feet. The Acute Mountain Sickness Symptom Scale and Score assessments will be conducted before breakfast and before sleep from arrival day to Day 3 after high altitude exposure. The difference will be compared in the mean Acute Mountain Sickness Symptom Scale and Score after arrival between Suxiao Jiuxin Pill and Placebo groups.
Rate of oxygen treatment after arrival between Suxiao Jiuxin Pill and Placebo groups. | Arrival day to Day 3 after high altitude exposure
  Oxygen treatment will be given according to the participants' requirement or care providers' suggestion. The difference will be compared in the rates of oxygen treatment after arrival between Suxiao Jiuxin Pill and Placebo groups.

OTHER OUTCOMES:
Change of blood pressure and heart rate at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups. | Baseline, Day 4 at sea level, arrival day, Day 3 after high altitude exposure
  Blood pressure and heart rate assessments will be conducted before breakfast, before lunch and before sleep at baseline and Day 4 at sea level, arrival day to Day 3 after high altitude exposure. The difference will be compared in the changes of blood pressure and heart rate at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups.
Change of brain natriuretic peptide (BNP) at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups. | Baseline, the next day after arrival, Day 3 after arrival
  BNP will be measured at baseline (at sea level), the next day after arrival and Day 3 after arrival. The difference will be compared in the changes of BNP at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups.
Change of pulmonary artery systolic pressure estimated by echocardiography at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups. | Baseline, the next day after arrival, Day 3 after arrival
  Pulmonary artery systolic pressure will be estimated by echocardiography at baseline (at sea level), the next day after arrival and Day 3 after arrival. The difference will be compared in the change of pulmonary artery systolic pressures at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups.
Rate of sleep disturbances at high altitude between Suxiao Jiuxin Pill and Placebo groups. | Baseline, Day 3 to Day 5 at sea level, the next day after arrival to Day 3 after arrival
  Sleep questionaires, including Athens Insomnia Scale and Epworth Sleepiness Scale, will be recorded at mornings of baseline, and Day 3 to Day 5 at sea level, and the next day after arrival to Day 3 after arrival. The difference will be compared in the rates of sleep disturbances at high altitude between Suxiao Jiuxin Pill and Placebo groups.
Change of carotid-femoral pulse wave velocity (cfPWV) at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups. | Baseline, the next day after arrival, Day 3 after arrival
  cfPWV will be measured at baseline (at sea level), the next day after arrival and Day 3 after arrival. The difference will be compared in the change of cfPWV at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups.
Change of mean velocity of middle cerebral artery at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups. | Baseline, the next day after arrival, Day 3 after arrival
  Mean velocity of middle cerebral artery will be measured using transcranial Doppler ultrasound at baseline (at sea level), the next day after arrival, and Day 3 after arrival. The difference will be compared in the changes of mean velocity of middle cerebral artery at high altitude from baseline between Suxiao Jiuxin Pill and Placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, M.D., Principal Investigator — Peking University First Hospital; Yan Zhang, M.D., Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No